CLINICAL TRIAL: NCT06771401
Title: Identification of Diagnostic, Prognostic and Predictive Biomarkers in Cervical Mucus for Reproductive and Gynecological Disorders
Brief Title: Identification of Biomarkers in Cervical Mucus
Acronym: IBISCUS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, SCAMBIA GIOVANNI, Professor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 7175
Record Dates: First submitted 2024-12-06; First posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Cervical Mucus Dysfunction; Infertility, Female
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CERVICAL MUCUS ANALYSIS (Other): Analysis of the characterization by infrared spectroscopy of cervical mucus and its variations during the different phases of the menstrual cycle in cases vs healthy controls groups
  Interventions: Diagnostic Test: cervical mucus sampling

INTERVENTIONS:
Diagnostic Test: cervical mucus sampling — Monitoring of menstrual cycle will be conducted in the follicular, ovulatory and luteal phases during which cervical mucus, serum and urine samples will be collected and pelvic ultrasound scans performed (3-5 ultrasound scans/samples within the cycle).

SUMMARY:
Cervical mucus is a biological fluid secreted by the endocervical glandular epithelium whose quantitative and qualitative characteristics vary in response to the hormonal stimulus produced by the ovary during the woman's menstrual cycle. As a fertility factor, it performs numerous biological functions: transport, nourishment, defense and capacitation of spermatozoa, defense against pathogens of the female genital tract.

The aim of this research will be to deepen the knowledge of the biochemical characteristics of cervical mucus, in particular to perform characterization by infrared spectroscopy, for the identification of diagnostic, prognostic and predictive biomarkers for disorders affecting the female reproductive system.

A healthy control population and a cohort of patients affected by unexplained infertility will be enrolled for the longitudinal study of the menstrual cycle with ultrasound and hormonal monitoring and serial sampling of cervical mucus.

ELIGIBILITY:
Inclusion Criteria:

* HEALTHY CONTROL

  * Women of 18-45 years old,
  * Use of the Billings Ovulation Method® for at least three months in the last three years
  * Proven fertility
* STUDY COHORT

  * Women of 18-45 years old,
  * Women affected by unexplained infertility

Exclusion Criteria:

* Virgo women
* Women incapable of understanding and wanting
* Women who have had sexual intercourse in the two days prior to cervical mucus sampling
* Pregnancy, exclusive breastfeeding
* Amenorrhea
* Gynecological hormone ongoing therapies or suspended for less than three months
* Cervico -vaginal infections
* Psychiatric pathologies
* Untreated/decompensated endocrine-metabolic disorders
* Coagulopathies and renal pathologies under dialysis treatment
* Refusal of informed consent
* Previous, current or suspected oncological pathology

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-01-10 (Estimated); Primary Completion 2026-07-10 (Estimated); Study Completion 2028-01-10 (Estimated)

PRIMARY OUTCOMES:
Characterization by infrared spectroscopy of cervical mucus | 1 month (3 time points within a menstrual cycle)
  Analysis of the spectra as revealed using by infrared spectroscopy on samples of cervical mucus. Analysis of their variations during the different phases of the menstrual cycle in cases group vs healthy controls groups.